CLINICAL TRIAL: NCT01397760
Title: Retrospective Study for Description of The Use Of Omalizumab In Patients With Difficult To Control Asthma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fiks, Iara Nely, M.D. (Individual)
Responsible Party: IARA NELY FIKS, IARA NELY FIKS
Other Study IDs: iara fiks 1
Record Dates: First submitted 2011-07-12; First posted 2011-07-20 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Asthma
Keywords: DIFFICULT TO CONTROL ASTHMA; OMALIZUMABE
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is do describe the experience in the use of omalizumabe, in a real life scenario, in uncontrolled severe asthmatic patients attended in specialist outpatient clinics, and its efficacy and safety. The efficacy of omalizumab in the population observed will be evaluated as reduction of uncontrolled asthma related events, i.e. exacerbations, emergency dept. visits, hospitalization and asthma-related treatment (decrease of asthma medication).

DETAILED DESCRIPTION:
Omalizumab is indicated in children over 6 years of age, with diagnosis of difficult to control asthma, presenting a component of atopy demonstrated preferably positive skin tests (prick test) or in vitro reactivity (rast) allergens common inhalants. Patients must also present the total serum IgE levels between 30 and 700UI/mL. Children until 12 years the IgE level is between 30 and 300 IU/ml.

ELIGIBILITY:
Inclusion Criteria:

Patients on optimal asthma treatment, good compliance and no response to treatment according to asthma consensus (GINA/NAEEP and the Latinamerican Consensus for Difficult to treat Asthma)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 PATIENTS WITH difficult to treat asthma
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Number of asthma hospitalization | ONE YEAR Of Omalizumab USE

SECONDARY OUTCOMES:
Decrease the doses of oral steroids | ONE YEAR Of Omalizumab USE

CONTACTS AND LOCATIONS:
Overall Officials: iara n fiks, md, Principal Investigator — pulmonary sao luiz hospital
Locations (1):
- Iara Nely Fiks, São Paulo, São Paulo, Brazil